CLINICAL TRIAL: NCT06150638
Title: Tratamiento de la distensión Abdominal Funcional Mediante Biofeedback no Instrumental
Brief Title: Treatment of Functional Abdominal Distension by Non-instrumental Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)459-2023
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome; Dyspepsia; Functional Bloating
MeSH Terms: conditions — Irritable Bowel Syndrome; Dyspepsia | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental)
  Interventions: Behavioral: Biofeedback
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Biofeedback — Three sessions of biofeedback intervention will be performed during the first 3 weeks of the intervention period. Patients will be taught to control abdominal and thoracic muscular activity by providing instructions using an original video support. Patients will be instructed to perform the same exercises before and after breakfast, lunch and dinner during the 4-week intervention period.
  Arms: Biofeedback
Behavioral: Placebo — Three sessions of placebo intervention will be performed during the first 3 weeks of the intervention period. Sham measurements of abdominal and thoracic motion will be performed, and a pill of placebo containing 0.21 g glucose will be administered; patients will be instructed to take a pill of placebo before breakfast, lunch and dinner during the 4-week intervention period.
  Arms: Placebo

SUMMARY:
Background. Abdominal distention is produced by an abnormal somatic postural tone. The authors developed an original biofeedback technique based on electromyography-guided control of abdominothoracic muscular activity. In a randomized, placebo-controlled trial the authors demonstrated the superiority of biofeedback over placebo for the treatment of abdominal distention. However, the technique is technically complex and unpractical.

Aim. To prove the efficacy of a non-instrumental biofeedback technique for the treatment of abdominal distension.

Selection criteria. Visible abdominal distension after meal ingestion; patients are able to identify the offending meal.

Intervention. Patients will be randomized into biofeedback in placebo groups. Three sessions of either biofeedback or placebo intervention will be performed during the first 3 weeks of the intervention period.

Biofeedback: patients will be taught to control abdominal and thoracic muscular activity by providing instructions using an original video support. Patients will be instructed to perform the same exercises before and after breakfast, lunch and dinner during the 4-week intervention period.

Placebo: sham measurements of abdominal and thoracic motion will be performed, and a pill of placebo containing 0.21 g glucose will be administered; patients will be instructed to take a pill of placebo before breakfast, lunch and dinner during the 4-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* episodes of visible abdominal distension triggered by meal ingestion
* patients are able to identify the offending foodstuff

Exclusion Criteria:

* organic cause detected by clinical work-up
* constipation
* abdominal distension not confirmed by the 7-day clinical questionnaires or after the probe meal in the pre-intervention evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Sensation of abdominal distension | 4 weeks
  Sensation score measured by scales graded from 0 (not at all) to 10 (very much) at the end of each day over a 7-day clinical evaluation period before and during the 4th week of the intervention.

SECONDARY OUTCOMES:
Changes in girth produced by the probe meal | 4 weeks
  Abdominal girth will be measured using a non-stretch belt that is placed over the umbilicus before and after the probe meal. The response to the meal will be measured before and after treatment.
Effect of probe meal on sensation of abdominal distension | 4 weeks
  Sensation score measured by scales graded from 0 (not at all) to 10 (very much) after the probe meal. The response to the meal will be measured before and after the intervention.

OTHER OUTCOMES:
Follow-up after biofeedback | 6 months
  Sensation of abdominal distension measured by scales graded from 0 (not at all) to 10 (very much) at the end of each day over a 7-day clinical evaluation period at 1, 3 and 6 months after biofeedback treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — University Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Barba E, Accarino A, Azpiroz F. Correction of Abdominal Distention by Biofeedback-Guided Control of Abdominothoracic Muscular Activity in a Randomized, Placebo-Controlled Trial. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1922-1929. doi: 10.1016/j.cgh.2017.06.052. Epub 2017 Jul 11. PMID 28705783